CLINICAL TRIAL: NCT00284973
Title: Ph-1 Double-Blind Randomized Control Study-Evaluate Safety & Immunogenicity of Wanxing Bio-Pharmaceuticals AMA-1/MSP-1 Recombinant Malaria Vaccine (PfCP-2.9) Adj. w/ Montanide ISA 720 Compared to Montanide ISA 720 Alone in Adult Volunteers
Brief Title: A Study of Safety and Immunogenicity of a Malaria Vaccine Candidate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Wanxing Bio-Pharmaceutical Co. Ltd. (Industry)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Second Military Medical University (Other); World Health Organization (Other); PATH (Other)
Organization: PATH (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WanMal002
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2007-04

CONDITIONS: Prophylaxis Against Plasmodium Falciparum Malaria
Keywords: malaria
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Biological: Plasmodium falciparum Chimeric Prot. 2.9 - Montanide ISA 720

SUMMARY:
Shanghai Wanxing Bio-Pharmaceuticals is currently evaluating one malaria vaccine candidate, PfCP2.9 adjuvanted with Montanide ISA 720. This trial is designed to test the safety and immunogenicity of 3 doses and 2 vaccination schedules.

This blood stage candidate malaria vaccine is being developed for the routine immunization of infants and children living in malaria-endemic areas.

DETAILED DESCRIPTION:
This is a double blind, randomized, controlled Phase I study of PfCp2.9, an experimental malaria vaccine candidate, adjuvanted with Montanide ISA 720.

The primary objective of this study is to assess the safety and reactogenicity of the vaccine in healthy Chinese adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female ≥ 18 and ≤ 45 years of age
* Agrees not to donate blood during the course of the trial.
* Signed written informed consent provided.
* Available to participate for the study duration.

Exclusion Criteria:

* History of allergic reactions following any vaccination.
* Involvement in drug or other vaccine trial within four weeks prior to the trial.
* Acute illness within four weeks prior to the trial.
* Presence of fever at the time of vaccination, i.e. body temperature (by axillary) > 37.5 C.
* Presence of any chronic illness/disease including diabetes mellitus, tuberculosis, leprosy, epilepsy and hypertension determined by medical history or examination.
* Persons on systemic corticosteroids, immunomodulators or anticoagulants within four weeks prior to vaccination.
* Persons with a history of allergic manifestations requiring treatment with injectable antihistamines, adrenaline or steroids.
* Pregnancy. Women should not be pregnant, lactating, or planning pregnancy throughout the study period. A urinary pregnancy test (immuno-chromatography) will be performed for all women of child-bearing potential at entry and prior to each vaccination. Adequate contraception throughout the study should be used if applicable.
* Sexually active woman not using contraceptives.
* Current smoker ( ≥ 20 cigarettes/day).
* History of malaria: persons with a known history of malaria or with positive markers for antibodies to malaria parasite by IFA and/or ELISA.
* History of residing in a malaria endemic region or malaria exposure (travel) within last two years.
* Abnormal hematology and clinical chemistry considered to be clinically significant.
* Abnormal urine routine test considered to be clinically significant
* Persons with positive markers for HBV (HBsAg) and/or HCV (Anti-HCV) infection.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70
Dates: Start 2006-01

PRIMARY OUTCOMES:
To assess the safety and reactogenicity of the PfCP-2.9 /Montanide ISA 720 vaccine in healthy adult volunteers.

SECONDARY OUTCOMES:
To assess the immunogenicity of the PfCP-2.9/Montanide ISA 720 vaccine in healthy adult volunteers by evaluating and comparing antigen-specific antibody responses (anti-PfCP-2.9 ELISA) after each vaccination.
For exploratory analysis:
To assess in vitro inhibition of parasite growth by vaccine-induced antibodies as measured by the GIA
To assess the relationship between antibody levels as measured by ELISA with the corresponding degree of in vitro parasite growth inhibition as measured by GIA
To assess antigen-specific antibody responses by IFA after each vaccination
To assess the relationship between antibody levels as measured by ELISA with IFA titers that recognize the conformational antigens of the parasite.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhong Hu, Dr., Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China